CLINICAL TRIAL: NCT04849169
Title: A Prospective, Multicenter, Single-arm Investigation of the Ringer Perfusion Balloon Catheter Performed Under an Exception From Informed Consent (EFIC) (Ringer IDE Study)
Brief Title: Investigation of the Ringer Perfusion Balloon Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ST3031
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental Arm (Experimental): Adult subjects who experience a perforation of a coronary vessel during percutaneous coronary intervention (PCI) and require management of hemorrhage until a definitive treatment is determined.
  Interventions: Device: Experimental

INTERVENTIONS:
Device: Experimental — Prolonged balloon inflation for hemorrhage management due to coronary artery perforation.

SUMMARY:
The objective of this study is to demonstrate reasonable assurance that the Ringer catheter can be safely used to manage hemorrhage due to coronary vessel perforations while facilitating distal perfusion under the conditions of use prescribed in the labeling.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm clinical study. The study will be conducted at up to 15 investigational sites in the US and will enroll up to 30 participants. The population for this investigation is adult participants who suffer a perforation of the coronary artery during a percutaneous coronary intervention requiring management of hemorrhage while providing distal perfusion until definite treatment is determined.

This clinical investigation is being conducted under Exception from Informed Consent (EFIC) regulations because there is no reasonable way to identify patients likely to become eligible for the investigation, and a coronary perforation can be a life-threatening emergency that needs to be immediately controlled without enough time for the patient or their legally authorized representative to give consent. Patients will be notified of their enrollment as soon as feasible. For more information on the exception from informed consent, please use the contact information be.ow.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of the PCI procedure
* Subject has fluoroscopically confirmed vessel perforation (classified as any type) requiring management of hemorrhage until a definitive treatment is determined
* Female subjects of childbearing potential must have a negative pregnancy test per standard of care for PCI

Exclusion Criteria:

-The perforation location prevents complete inflation or proper placement of the Ringer catheter, as detailed in the Instructions for Use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness of device success in managing hemorrhage while preserving flow | Procedure
  Effectiveness of device success in managing hemorrhage while preserving flow via angiographic confirmation of: a) successful delivery of Ringer across perforation, b) acute cessation of extravasation while Ringer is inflated, and c) demonstration of antegrade blood flow during Ringer deployment.
Rate of Ringer related thrombosis and/or dissection | Procedure
  Rate of Ringer-related thrombosis and new or worsening coronary dissection following Ringer deflation and withdrawal.

SECONDARY OUTCOMES:
Change in TIMI (thrombolysis in myocardial infarction) flow | Procedure
  The change in TIMI flow during Ringer deployment.
Change in perforation classification | Procedure
  The change in perforation classification after Ringer deployment
Rate of clinically relevant events | Discharge or 30 days, whichever comes first.
  Rate of clinically relevant events in the management of the coronary perforation and any potential sequelae including: chest pain, bleeding incidence and severity, major adverse cardiac events (MACE), cardiac tamponade and pericardiocentesis, emergency surgery post-perforation including coronary artery bypass graft (CABG), death.

CONTACTS AND LOCATIONS:
Overall Officials: David E Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (6):
- United States (6):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory Heart & Vascular Center, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No